CLINICAL TRIAL: NCT06009055
Title: Effects of Remimazolam and Propofol on Heart Rate Variability in Type 2 Diabetes Patients During Anesthesia Induction
Brief Title: Effects of Remimazolam and Propofol on Anesthesia Induction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zheng Guo (Other)
Responsible Party: Sponsor-Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Organization: Second Hospital of Shanxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hanyi20230117
Record Dates: First submitted 2023-02-17; First posted 2023-08-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental)
  Interventions: Drug: Remimazolam
- Propofol group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — 0.3mg/kg，injection completed in 30 seconds
  Arms: Remimazolam group
Drug: Propofol — 2mg/kg，injection completed in 30 seconds
  Arms: Propofol group

SUMMARY:
The patients with diabetes who underwent laparoscopic cholecystectomy in the general surgery department of the Second Hospital of Shanxi Medical University were selected. The patients who were induced by remimazolam were included in the experimental group, and the patients who were induced by propofol were included in the control group. All the selected patients had no intimate relationship. The differences of blood pressure, heart rate and heart rate variability (HRV) between the experimental group and the control group were observed. According to the literature, it is speculated that the changes of blood pressure, heart rate and HRV indexes in the experimental group are smaller than those in the control group, and the difference is statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as type 2 diabetes according to the "Chinese Guidelines for the Prevention and Treatment of Type 2 diabetes 2020"
* ASA II or III

Exclusion Criteria:

* People who are allergic to Remimazolam
* It is estimated that patients with difficulty in tracheal intubation (poor head and neck mobility, history of airway surgery, history of OSAHS, nail to chin distance<6cm, Malampati grade 3 and above, mouth opening<2.5cm, obesity (BMI>30kg · m-2), etc
* Hypertension (clinically diagnosed as hypertension)
* Patients with coronary heart disease (with typical symptoms of angina pectoris and exclusion of aortic valve disease, clear history of old myocardial infarction, clear history of acute myocardial infarction, coronary stenosis greater than or equal to 70% found by CAG)
* Patients with arrhythmia, heart failure, renal failure, and recently taking cardiovascular active drugs
* Endocrine diseases such as hyperthyroidism and pheochromocytoma that may affect the level of body hemodynamics
* Ketoacidosis and lactic acidosis
* Patients with long-term use of sedatives or antidepressants or a history of alcoholism or drug dependence
* Asthma or reactive airway disease
* Patients with myasthenia gravis and cognitive dysfunction cannot cooperate with this study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
systolic pressure （SBP） | 24 hours
  Changes in systolic blood pressure
diastolic pressure（DBP） | 24 hours
  change of diastolic blood pressure
heart rate | 24 hours
  change of heart rate
Heart rate variability（HRV） | 24 hours
  Changes of various indicators of heart rate variability

CONTACTS AND LOCATIONS:
Locations (1):
- econd of Shanxi Medical University, Taiyuan, Shanxi, China